CLINICAL TRIAL: NCT03726853
Title: A Phase 2, Randomized, Double-blind, Multi-center, Parallel-group Trial to Evaluate the Efficacy and Safety of CKD-497
Brief Title: The Clinical Trial to Evaluate the Efficacy and Safety of CKD-497
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 176AURI/AB17014
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2018-11

CONDITIONS: Respiratory Infection
Keywords: Acute upper respiratory infection; Acute bronchitis
MeSH Terms: conditions — Respiratory Tract Infections; Bronchitis | interventions — CKD-497

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CKD-497 200mg (Experimental): CKD-497 200mg
  Interventions: Drug: CKD-497 200mg; Drug: Comparator placebo
- CKD-497 300mg (Experimental): CKD-497 300mg
  Interventions: Drug: CKD-497 300mg; Drug: Comparator placebo
- Active Comparator (Active Comparator): compartor
  Interventions: Drug: CKD-497 placebo; Drug: Comparator
- Placebo (Placebo Comparator): CKD-497 placebo and comparator placebo
  Interventions: Drug: CKD-497 placebo; Drug: Comparator placebo

INTERVENTIONS:
Drug: CKD-497 200mg — CKD-497 200mg
  Arms: CKD-497 200mg
Drug: CKD-497 300mg — CKD-497 300mg
  Arms: CKD-497 300mg
Drug: CKD-497 placebo — Placebo of CKD-497
  Arms: Active Comparator; Placebo
Drug: Comparator — Comparator
  Arms: Active Comparator
Drug: Comparator placebo — Comparator placebo
  Arms: CKD-497 200mg; CKD-497 300mg; Placebo

SUMMARY:
To evaluate the efficacy and safety of CKD-497

ELIGIBILITY:
Inclusion Criteria:

1. 19 ≤ age < 75
2. Subject with acute upper respiratory infection and acute bronchitis infection
3. Subject who agreeds to participate in this clinical trial voluntarily

Exclusion Criteria:

1. Subject who need antibiotics treatment during the clinical trial
2. Subject suffering from severe respiratory diseases such as pneumonia, asthma, chronic closed lung diseases (COPD), tuberculosis, bronchial enlargement, malignant tumors in the lungs, and chronic bronchitis during screening
3. Subject who cannot participate in a clinical trial based on the PI's judgment

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
BSS(Bronchitis Severity Score) | 1 week
  0(absent) ~ 4(very severe), Total Score: 0~20
SUM8(The 8-symptom related questions in the Daily Cough and Phlegm) | 1 week
  0(Never) ~ 4(always), Total Score: 0~32

CONTACTS AND LOCATIONS:
Locations (15):
- South Korea (15):
  - Ulsan University Hospital, Ulsan, Dong-gu
  - KyungHee University Medical Center, Seoul, Dongdaemun-gu
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, Dongjak-gu
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Konkuk University Medical Center, Seoul, Gwangjin-gu
  - Hanyang University Guri Hospital, Guri-si, Gyenggi-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Kangbuk Samsung Hospital, Seoul, Jongno-gu
  - Kangdong Sacred Heart Hospital, Seoul, Kangdong-gu
  - Gachon University Gil Medical Center, Incheon, Namdong-gu
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul, Seocho-gu
  - Korea University Anam hospital, Seoul, Seongbuk-gu
  - EWHA Womans University Mokdong Hospital, Seoul, Yangcheon-gu
  - The Catholic University of Korea, Yeouido ST. Mary's Hospital, Seoul, Yeongdeungpo-gu

IPD SHARING:
Plan to Share IPD: No